CLINICAL TRIAL: NCT00159185
Title: Epidemiology Study in Major Orthopaedic Surgery
Status: Completed | Type: Observational
Sponsor: Hoersholm Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: ESMOS
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-09

CONDITIONS: Thrombosis; Postoperative Complications; Quality of Life
Keywords: Arthroplasty, Replacement, Hip; Epidemiology
MeSH Terms: conditions — Thrombosis; Postoperative Complications

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to:

* Create a database including a description of the patient population that undergoes total hip replacement with special emphasis on orthopedic and cardiovascular complications and the quality of life 1 year postoperatively.
* Characterise the patient at risk for the above mentioned events
* Create methods for predicting patients at risk for short-term (90 days) and long term (1 year) complications in relation to hip replacement surgery.

DETAILED DESCRIPTION:
Introduction:

Total hip replacement surgery is a standard procedure, which has been shown to be both cost-effective and to give the patient a pain free daily living. Since Sir Charnley made total hip replacement a standard procedure millions of hips have been implanted.

In Denmark about 100 out of 100.000 did get a hip replacement operation in 2001(DHAR).

When a patient with a painful hip due to arthrosis, arthritis, fracture sequelae and other reasons, is offered a total hip replacement, several issues are taken into consideration: concurrent diseases, bone quality, age, life expectancy, prosthesis type, operation methods etc.

In the elderly patient a thorough medical evaluation is performed in order to minimise the intraoperative risc for cardiopulmonary morbidity. Nearly all patients in Denmark (over 99%) are getting thromboprophylaxis during the hospital stay to minimise cardiovascular complications.

After surgery the patients visits the outpatient clinic for routine control after 3 and 12 months. After that time the patient is usually out of orthopedic control.

Evaluations of the procedures in Scandinavian countries are collected in databases. These databases are constructed by national collection of data sheets from each hospital performing the procedures. The collected data most often only include data as far as the arthroplasty is concerned. Normally there is no monitoring of the quality of the collected data - a considerable margin of errors in the results produced from these databases must there for be expected.

The amount of publications concerning total joint replacement is enormous, but most publications in this field come from clinical trials dealing with new pharmacological products or new implants.

Very few authors have considered the overall patient morbidity and quality of life after the hip replacement operation.

Therefore this Ph.D. project is planned to get more and newer data of the population that is offered a total hip replacement. Furthermore, it will be attempted to find prognostic factors as far as the overall risk for cardiopulmonary complications in the first 1 - 3 years after the operation.

Purpose:

The purpose of this study is to:

Create a database including a description of the patient population that undergo total hip replacement with special emphasis on orthopedic and cardiovascular complications and the quality of life 1 year postoperatively.

Characterise the patient at risk for the above mentioned events

Create methods for predicting patients at risk for short-term (90 days) and long term (1 years) complications in relation to hip replacement surgery.

Hypothesis:

It is a well defined small group of high risk patients that gets the serious cardiovascular complications.

The risk for cardiovascular complications is increased for a longer period than the postoperative hospital stay.

A not neglectable group of the patients do not get the expected benefit from the operation.

Methods:

A prospective monocentre, longitudinal cohort study of 500 patients operated in the County of Frederiksborg from 01.01 2004.

The data will be collected by interview before the operation, on day 5 and after 3 month and a year.

And additional data will be collected from patient files, local hip- and anaesthesia databases, laboratory system, the Danish Hospital Discharge Register (LPR), autopsy reports and death register.

Statistical methods:

In the PhD study is included various courses, including a course on statistical methods. External statistical aid might be necessary.

Patients:

Inclusion criteria:

All patients to be operated with total hip replacement in Frederiksborg amt from 01.01.2004 until 500 pt. have been included.

Exclusion criteria:

Refuse of consent and age under 18years.

Ethical Considerations:

Local Scientific Ethical Committee and theDanish Dataprotection Agency has to approve the project.

The project follows the Guidelines for Good Clinical Practise.

The investigation will not imply any discomfort and no risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated with Hip Arthroplasty Replacement in Hillerød and Hørsholm Hospitals from 1.1 2004.

Exclusion Criteria:

* Written informed consent denied
* Patients under 18 years of age.
* Patients not habitants of Denmark at the time of the operation.
* Patients without a CPR-number (civil registration number).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-01; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Ryge, MD, Study Chair — Hoersholm Hospital
Locations (1):
- Hoersholm Hospital, Hoersholm, Hoersholm, Denmark